CLINICAL TRIAL: NCT03157830
Title: Evaluating the Efficacy and Safety of Transitioning Patients From Natalizumab to Ocrelizumab
Acronym: OCTAVE
Status: Completed | Type: Observational
Sponsor: Providence Health & Services (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39655
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; ocrelizumab; OCREVUS; Natalizumab; Tysabri
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Ocrelizumab, OCREVUS: Patients eligible for this study will be receiving OCREVUS as part of their routine care for MS treatment, and undergo the standard monitoring tests and procedures for MS patients receiving treatment. In addition, they will complete the EDSS scale on 6 occasions over a 12-month period, and the MSIS-29 on three occasions during the 12 month period for research.

SUMMARY:
The primary objective of this study is to assess the efficacy of Ocrelizumab (OCR) in Relapsing Multiple Sclerosis patients who have been previously treated with natalizumab (NTZ) by evaluating relapse rate, progression on MRI and disability progression.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label, Phase IV clinical trial. Patients with relapsing forms of Multiple Sclerosis (MS), ages 18 to 65, who have received a stable dose of NTZ for 12 or more consecutive months, and have been free of relapses, disability worsening or Magnetic Resonance Imaging (MRI) progression 6 months prior to the transition screening visit will be eligible for the study. After informed consent to participate has been obtained, the patient will have physical exam (PE), non-blinded Expanded Disability Status Scale (EDSS), MRI, Multiple Sclerosis Impact Scale (MSIS-29) and labs done for the screening visit to determine eligibility. Brain MRI with and without contrast will be performed with the standard MS protocol. MRIs will be performed with 3mm slice thickness with no gaps between slices. Patients will receive their first dose of OCR 4 to 6 weeks after the last dose of NTZ. Other baseline measures, including physical exam, EDSS, MSIS-29, and labs will be performed within 4 weeks of screening. Physical exam, non-blinded EDSS, and labs will be performed at month 3, month 6, month 9, and month 12. MSIS-29 will be performed at months 6 and 12. In addition, MRIs will be performed at months 3, 6, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with relapsing form of MS, age 18 to 65, inclusive, at the time of informed consent.
* In the opinion of the investigator, able to understand the purpose and risk of the study and provide signed informed consent document.
* Must have received a stable dose of NTZ for 12 or more consecutive months, and have had no evidence of on-NTZ disease activity (clinically or on MRI) for the 6 months prior to the screening visit.
* Naïve to OCR.
* No evidence, in the opinion of the investigators of significant cognitive limitation or psychiatric disorder that would interfere with the conduct of the study.
* EDSS of ≤ 6.0 at screening.
* Female patients of childbearing potential must practice effective contraception and continue contraception during the study.

Exclusion Criteria:

* History of primary or secondary progressive multiple sclerosis.
* Evidence of active hepatitis B infection at screening.
* Any mental condition of such that patient is unable to understand the nature, scope, and possible consequences of the study.
* Patients with untreated hepatitis C or tuberculosis. Patients who have history of progressive multifocal leukoencephalopathy (PML) or known to be HIV positive, per standard care.
* Any persistent or severe infection.
* Pregnancy or lactation.
* Significant or uncontrolled somatic disease or severe depression in the last year.
* Inability to complete an MRI.
* Previous treatment with B-cell targeted therapies.
* Current use of immunosuppressive medication.
* Patients who have had evidence of disease activity within the 6 months prior to screening. This includes MS relapse, or new or enlarging T2 lesions or Gd+ enhancing lesions, or disability progression.
* Patients with any significant comorbidity that in the opinion of the investigator, would interfere with participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with relapsing forms of MS, ages 18 to 65, must have received a stable dose of NTZ for 12 or more consecutive months, and have been free of relapses, disability worsening or MRI progression 6 months prior to switching from NTZ to OCR therapy are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Smoot, MD, Principal Investigator — Providence Brain & Spine Institute
Locations (5):
- United States (5):
  - RWJBarnabas Health, Livingston, New Jersey
  - Providence MS Center, Portland, Oregon
  - Kadlec Neuroscience Center, Richland, Washington
  - Multiple Sclerosis Center, Swedish Neuroscience Institute, Seattle, Washington
  - Providence Multiple Sclerosis Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smoot K, Marginean H, Gervasi-Follmar T, Chen C, Repovic P, Cohan S. Evaluating the efficacy and safety of transitioning patients with multiple sclerosis from natalizumab to ocrelizumab (OCTAVE). Mult Scler. 2023 Jul;29(8):956-966. doi: 10.1177/13524585231175284. Epub 2023 Jun 15. PMID 37317841
- See also: Providence Brain & Spine Institute — http://oregon.providence.org/our-services/p/providence-brain-and-spine-institute/?utm_source=bing&utm_medium=cpc&utm_campaign=Brand%20-%20PBSI&utm_term=%2Bprovidence%20%2Bbrain%20and%20%2Bspine%20%2Binstitute&utm_content=PBSI_BMM&gclid=CNHRxL728tMCFSUhfgodHSsOHg&gclsrc=ds&dclid=CPq-0r728tMCFZGEYgod7ZgOAw

RESULTS

PARTICIPANT FLOW:
Groups:
- Ocrelizumab, OCREVUS: Patients eligible for this study will be receiving OCREVUS (also known as Ocrelizumab) as part of their routine care for multiple sclerosis (MS) treatment, and undergo the standard monitoring tests and procedures for multiple sclerosis (MS) patients receiving treatment. In addition, they will complete the Expanded Disability Status Scale (EDSS) scale on 6 occasions over a 12-month period, and the Multiple Sclerosis Impact Scale (MSIS-29) on three occasions during the 12 month period for research.
Period: Overall Study
Arm/Group | Ocrelizumab, OCREVUS
Started | 43
Completed | 41
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 43
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 43 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 2
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 43
Disease duration [Median (Inter-Quartile Range); unit: Years] | 11 [1 to 29]

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival at Month 12
Description: The proportion of relapse-free patients at month 12 after switching from natalizumab to ocrelizumab.
Time Frame: 12 Months
Measure: Number (95% Confidence Interval); unit: Percentage of Participant Survival Rate
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 43
Percentage of Participant Survival Rate | 95.2 [88.9 to 100]

2. Secondary Outcome: Relapse Rate at Months 3, 6, and 9
Description: Proportion of relapse-free patients at months 3, 6, and 9
Time Frame: 3, 6, and 9 months
Measure: Number; unit: percentage of relapse-free patients
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 43
percentage of relapse-free patients
  Proportion of relapse-free patients at months 3 | 100
  Proportion of relapse-free patients at months 6 | 100
  Proportion of relapse-free patients at months 9 | 97.67

3. Secondary Outcome: MRI Evidence of MS Disease Activity at Months 3, 6, and 12
Description: Proportion of patients free from MRI evidence of MS disease activity at months 3, 6, and 12
Time Frame: 3, 6, and 12 Months
Population: Number analyzed in one or more rows differs from overall number analyzed due to patients withdrawing prior to MRI scans at month 3. Additionally two patients showed evidence of MRI activity prior to MRI scans.
Measure: Number; unit: percentage of patients free from MRI evi
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 41
percentage of patients free from MRI evi
  Proportion of patients free from MRI evidence of MS disease activity at 3 months: number analyzed (Participants) | 39
  Proportion of patients free from MRI evidence of MS disease activity at 3 months | 92.31
  Proportion of patients free from MRI evidence of MS disease activity at 6 months: number analyzed (Participants) | 39
  Proportion of patients free from MRI evidence of MS disease activity at 6 months | 92.31
  Proportion of patients free from MRI evidence of MS disease activity at 12 months: number analyzed (Participants) | 39
  Proportion of patients free from MRI evidence of MS disease activity at 12 months | 92.31

4. Secondary Outcome: New or Enlarging T2 Lesions at 3, 6, and 12 Months
Description: Proportion of patients with New or Enlarging T2 lesions at 3, 6, and 12 months. For patients with New or Enlarging T2 lesions, number of New and Enlarging T2 lesions.
Time Frame: 3, 6, and 12 months
Measure: Number; unit: percentage of participants with new or e
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 43
percentage of participants with new or e
  Proportion of participants with new or enlarging T1 and/or T2 lesions at 3 months | 4.65
  Proportion of participants with new or enlarging T1 and/or T2 lesions at 6 months | 0
  Proportion of participants with new or enlarging T1 and/or T2 lesions at 12 months | 0

5. Secondary Outcome: New Gd+ Lesions Detected at Months 3, 6, and 12
Description: Proportion of patients with New Gd+ lesions detected at months 3, 6, and 12. For patients with New Gd+ lesions, number of New Gd+ lesions
Time Frame: 3, 6, and 12 months
Measure: Number; unit: percentage of participants with new Gd+
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 39
percentage of participants with new Gd+
  Proportion of patients with new Gd+ lesions at 3 months | 5.13
  Proportion of patients with new Gd+ lesions at 6 months | 0
  Proportion of patients with new Gd+ lesions at 12 months | 0

6. Secondary Outcome: Change in the EDSS Score From Baseline to Month 12
Description: Average change in EDSS score. The Expanded Disability Status Scale (EDSS) is an assessment used by neurologist to assess changes in the level of disability over time in patients with MS. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scores are also based on measures of impairment in the 8 functional systems. Higher scores indicate greater impact of MS on QoL.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: Score on EDSS
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 43
Score on EDSS
  Baseline | 3.50 [1 to 6]
  Month 12 | 3.50 [1 to 6.5]

7. Secondary Outcome: Change in MSIS-29 From Baseline to Months 6 and 12
Description: Average change in MSIS-29: Multiple Sclerosis Impact Scale (MSIS) is a patient reported outcome (PRO) measure, consisting of two subscales- physical impact of MS (20 items) and psychological impact (9 items). It asks subject to rate the impact MS has their daily life in the past 2 weeks (1=low impact to 4=large impact). Scores from individual items are summed to a total score. Physical impact score ranges from 20-80 and psychological impact scores ranges from 9-36.
  Higher scores indicate greater impact of MS on QoL.
Time Frame: 6 and 12 months
Measure: Median (95% Confidence Interval); unit: score on MSIS29 Scale
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 43
score on MSIS29 Scale
  Physical - Baseline to Month 6 | -1.346 [-1.763 to 4.455]
  Psychological - Baseline to Month 6 | -1.283 [-2.086 to 0.4455]
  Physical - Baseline to Month 12 | 1.524 [-5.085 to 2.036]
  Psychological - Baseline to Month 12 | -0.6953 [-3.225 to 4.616]

8. Secondary Outcome: Proportion of Patients That Discontinued OCR
Description: Proportion of patients that stop treatment with OCR for any reason
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Ocrelizumab, OCREVUS
Number analyzed (Participants) | 43
percentage of participants | 4.65

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Ocrelizumab, OCREVUS
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 8/43
Other Adverse Events (participants affected / at risk) | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab, OCREVUS (N=43)
Urinary tract infection (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Spontaneous abortion (Reproductive system and breast disorders) | 1 (1)
Chronic venous hypertension with symptomatic varicose veins, left leg (Vascular disorders) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Acute encephalopathy (Immune system disorders) | 1 (1)
Acute cystitis without hematuria (Renal and urinary disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Malignancy, right breast* (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab, OCREVUS (N=43)
Infusion related reaction (General disorders) | 31 (31) — Treatment Related Adverse Event
Respiratory tract infection (Infections and infestations) | 12 (12) — Treatment Related Adverse Event
Urinary tract infection (Infections and infestations) | 7 (7) — Treatment Related Adverse Event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT03157830/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03157830/ICF_001.pdf